CLINICAL TRIAL: NCT01392430
Title: Discontinuation of Primary and Secondary Prophylaxis for Opportunistic Infections in HIV-infected Patients Who Had CD4+ Cell Count <200 Cells/mm3 But Undetectable Plasma HIV-1 RNA
Brief Title: Discontinuation of Primary and Secondary Prophylaxis for Opportunistic Infections in HIV-infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Romanee Chaiwarith, Faculty of Medicine, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OI prophylaxis
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: HIV Infection
Keywords: Primary prophylaxis; Secondary prophylaxis; Discontinuation
MeSH Terms: conditions — HIV Infections | interventions — Dapsone; Fluconazole; Itraconazole; Azithromycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (No Intervention): Continuation of prophylaxis of opportunistic infections
- Arm B (Experimental): Discontinuation of opportunistic infections
  Interventions: Other: Discontinuation of prophylactic drugs i.e. co-trimoxazole, dapsone, fluconazole, itraconazole, azithromycin

INTERVENTIONS:
Other: Discontinuation of prophylactic drugs i.e. co-trimoxazole, dapsone, fluconazole, itraconazole, azithromycin — Discontinuation of prophylaxis for opportunistic infections
  Arms: Arm B

SUMMARY:
The purpose of this study is to compare the incidence of opportunistic infections between HIV-infected patients who continue and discontinue primary or secondary prophylaxis for opportunistic infections in whom receiving combination antiretroviral therapy and achieve undetectable HIV-1 RNA, but CD4 cell counts are less than 200 cells/mm3.

DETAILED DESCRIPTION:
Currently, combination antiretroviral therapy (cART) has become the standard of care in the treatment of HIV infection in many parts of the world including Thailand. The benefits of cART represented by an increment of CD4 cell count and a suppression of HIV viral load have been reported worldwide. The National Institute of Health (NIH), the Centers for Disease Control and Prevention (CDC), and the HIV Medicine Association of the Infectious Diseases Society of America (HIVMA/IDSA) recommended discontinuing primary and secondary prophylaxis for prevention of opportunistic infections (OIs) in HIV-infected adults and adolescents receiving cART, when the CD4 cell count increase to a certain level for a certain period of time. For instances, Pneumocystis jiroveci pneumonia (PCP) prophylaxis can be discontinued when patients receiving HAART and CD4 ≥ 200 cells/mm3 for at least 3 months (for primary prophylaxis) or at least 6 months (for secondary prophylaxis), prophylaxis for Cryptococcal meningitis, disseminated penicilliosis, cerebral toxoplasmosis, and disseminated mycobacterium avium complex can be discontinued when patients receiving HAART and CD4 ≥ 100 cells/mm3 for at least 6 months. Our practices follow this guideline. However, recently there are new data showing that there were no cases developed PCP after primary or secondary prophylaxis discontinuation even if CD4 cell count < 200 cells/mm3. Discontinuation of secondary prophylaxis resulted in reduction in pill burdens that may improve HAART adherence, decrease drug-drug interactions, and also prevent drug adverse events that may happen.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. regularly receiving highly active antiretroviral therapy (HAART) during follow up
3. CD4 cell count < 200 cells/mm3
4. HIV-1 RNA < 50 copies/ml after receiving HAART
5. receiving primary or secondary prophylaxis for opportunistic infections including infections caused by Pneumocystis jiroveci, Cryptococcus neoformans, Penicilliosis marneffei, Histoplasma capsulatum, Toxoplasma gondii, Mycobacterium avium complex
6. given written informed consent

Exclusion Criteria:

1) pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Incidence of opportunistic infections | Participants will be followed up to 135 weeks
  To test whether the incidence of opportunistic infections differs between these 2 groups
  * Patients receiving cART and discontinue primary or secondary prophylaxis if their HIV-1 RNA achieve undetectable level.
  * Patients receiving cART and continue primary or secondary prophylaxis even if HIV-1 RNA achieve undetectable level.

CONTACTS AND LOCATIONS:
Overall Officials: Romanee Chaiwarith, MD, MHS., Principal Investigator — Maharaj Nakorn Chiang Mai Hospital, Department of Medicine, Chiang Mai University
Locations (1):
- Maharaj Nakorn Chiang Mai Hospital, Department of Medicine, Chiang Mai University, Muang, Chiang Mai, Thailand

REFERENCES:
- [Derived] Chaiwarith R, Praparattanapan J, Nuntachit N, Kotarathitithum W, Supparatpinyo K. Discontinuation of primary and secondary prophylaxis for opportunistic infections in HIV-infected patients who had CD4+ cell count <200 cells/mm(3) but undetectable plasma HIV-1 RNA: an open-label randomized controlled trial. AIDS Patient Care STDS. 2013 Feb;27(2):71-6. doi: 10.1089/apc.2012.0303. PMID 23373662